CLINICAL TRIAL: NCT00461006
Title: A Randomized, Double Blind Study to Compare the Effects of Aleglitazar and Actos on Glomerular Filtration Rate and Other Parameters of Renal Function in Patients With Type 2 Diabetes.
Brief Title: A Comparison of the Effects of Aleglitazar and Actos on Renal Function on Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC20653
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aleglitazar (Experimental)
  Interventions: Drug: aleglitazar
- Actos (Active Comparator)
  Interventions: Drug: Actos

INTERVENTIONS:
Drug: Actos — 45mg po daily
  Arms: Actos
Drug: aleglitazar — 0.6mg po daily
  Arms: Aleglitazar

SUMMARY:
This 2 arm study will compare the effects of aleglitazar and Actos, added to preexisting oral antihyperglycemic therapy and/or diet and exercise, on renal function in patients with type 2 diabetes, and normal or mildly impaired renal function. Eligible patients will be randomized to receive either aleglitazar 0.6mg p.o. or Actos 45mg p.o. daily. Renal function and efficacy parameters will be assessed at intervals during the treatment period. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes for >=1 month;
* drug naive, or receiving stable oral antihyperglycemic medication;
* HbA1c 6.5-10.0% at screening.

Exclusion Criteria:

* type 1 diabetes;
* current or previous treatment with insulin;
* history of renal disease other than diabetic nephropathy;
* uncontrolled hypertension;
* clinically significant cardiovascular disease;
* Congestive heart failure (CHF) New York Heart Association (NYHA) 3-4.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in glomerular filtration rate | 26 weeks

SECONDARY OUTCOMES:
Relative change from baseline in estimated renal plasma flow (ERPF) and urine albumin-creatinine ratio (UACR) | 26 weeks
Absolute change in Hemoglobin A1c (HbA1c), fasting plasma glucose (FPG) and fasting plasma insulin (FPI). | End of treatment
Adverse events (AEs), laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- United States (15):
  - Peoria, Arizona
  - Jonesboro, Arkansas
  - Fresno, California
  - Los Gatos, California
  - Mission Viejo, California
  - Jacksonville, Florida
  - Omaha, Nebraska
  - Charlotte, North Carolina
  - Marion, Ohio
  - Altoona, Pennsylvania
  - Arlington, Texas
  - Dallas, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
- Mexico (6):
  - Chihuahua City
  - Hermosillo
  - Metepec
  - Mexico City
  - Monterrey
  - Zapopan
- Puerto Rico (3):
  - Manatí
  - Ponce
  - Toa Baja
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Saratov
  - Tyumen
  - Yaroslavl
- Ukraine (7):
  - Dnipro
  - Donetsk
  - Kharkiv
  - Kiev
  - Lugnansk
  - Poltava
  - Ternopil